CLINICAL TRIAL: NCT00085293
Title: Phase II Study of Decitabine in Patients With Metastatic Papillary Thyroid Cancer or Follicular Thyroid Cancer Unresponsive to Radioiodine
Brief Title: Decitabine in Treating Patients With Metastatic Papillary Thyroid Cancer or Follicular Thyroid Cancer Unresponsive to Iodine I 131
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00033; NCI-2009-00033 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000368467; 5954; 2003-0308 (Other: M D Anderson Cancer Center); 5954 (Other: CTEP); P30CA016672 (NIH); N01CM62207 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Thyroid Cancer; Stage IVA Follicular Thyroid Cancer; Stage IVA Papillary Thyroid Cancer; Stage IVB Follicular Thyroid Cancer; Stage IVB Papillary Thyroid Cancer; Stage IVC Follicular Thyroid Cancer; Stage IVC Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Decitabine; Iodine-131; Thyrotropin Alfa; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Starting dose 6 mg/m^2 Decitabine intravenous (IV) over 1 hour on days 1-5 and 8-12 of weeks 1 and 2 (course 1). Week 3, Iodine I 131 (131I) scanning using thyrotropin alfa injections. Participants whose scan do not demonstrate iodine uptake continue suppressive thyroid hormone therapy but no further study therapy; these participants who do show uptake undergo thyroid hormone withdrawal on weeks 4-8 and second course of decitabine (as in course 1) on weeks 7 and 8, with 131I therapy on week 9.
  Interventions: Drug: Decitabine; Radiation: Iodine I 131; Biological: Recombinant thyrotropin alfa; Radiation: Fludeoxyglucose F 18; Procedure: Positron emission tomography

INTERVENTIONS:
Drug: Decitabine — Starting dose 6 mg/m^2 intravenously over 1 hour every day for 5 successive days for 2 weeks (10 doses), with possible second course.
  Other Names: 5-aza-dCyd; 5AZA; DAC
Radiation: Iodine I 131 — Undergo thyrotropin-alfa stimulated radioactive iodine scan
  Other Names: I 131; Iodotope; Iodotrope
Biological: Recombinant thyrotropin alfa — Undergo thyrotropin-alfa stimulated radioactive iodine scan
  Other Names: Thyrogen
Radiation: Fludeoxyglucose F 18 — Optional correlative studies
  Other Names: 18FDG; FDG
Procedure: Positron emission tomography — Optional correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase II trial is studying how well decitabine works in treating patients with metastatic papillary thyroid cancer or follicular thyroid cancer that has stopped responding to radioactive iodine. Iodine I 131 (radioactive iodine) kills thyroid cancer cells. Metastatic thyroid cancer cells can lose the ability to be treated with radioactive iodine. Decitabine may help thyroid cancer cells regain the ability to respond to treatment with radioactive iodine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether decitabine can restore iodine I 131 (131I) uptake in patients with metastatic papillary thyroid or follicular thyroid cancer lesions that are undetectable by low-dose iodine 131I scanning.

SECONDARY OBJECTIVES:

I. Determine the efficacy of 131I therapy, administered after restoration of 131I uptake by decitabine, in these patients.

II. Determine the effect of decitabine on clinical and molecular markers of thyroid cancer cell differentiation in these patients.

III. Determine the safety and tolerability of decitabine in patients undergoing thyroid hormone withdrawal-induced hypothyroidism and 131I therapy.

OUTLINE: This is an open-label, multicenter study.

Patients receive decitabine intravenous (IV) over 1 hour on days 1-5 and 8-12 of weeks 1 and 2 (course 1). On week 3, patients undergo iodine I 131 (131I) scanning using thyrotropin alfa injections. Patients whose scan does not demonstrate iodine uptake continue suppressive thyroid hormone therapy but receive no further study therapy. These patients undergo study follow up.

Patients whose scan demonstrates iodine uptake undergo thyroid hormone withdrawal on weeks 4-8 and receive a second course of decitabine (as in course 1) on weeks 7 and 8. Patients then receive 131I therapy on week 9.

Patients are followed at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed papillary thyroid or follicular thyroid carcinoma:

  * Differentiated disease;

    * Metastatic disease documented by ultrasound, computed tomography (CT) scan (without iodinated contrast), or MRI - All metastatic disease foci =< 10 mm in all dimensions
* Must have been treated with total or near-total thyroidectomy AND at least 1 course of iodine I 131 (131I)(>=29.9 mCi) OR demonstrated negative uptake on a postoperative low-dose131I scan
* Must have undergone whole body 131I scan 1-3 days after administration of =< 5.5 mCi of 131I demonstrating no visible iodine uptake within the lesions unless demonstrated negative uptake on a postoperative low-dose131I scan within the past 12 weeks:

  * Must have 24-hour urine iodine excretion =< 500 mcg within 1 week of 131I scan
* Must be receiving thyroid hormone therapy AND have thyroid-stimulating hormone level =< 0.5 mU/L
* No known brain metastases
* Performance status:

  * Eastern Cooperative Oncology Group (ECOG) 0-2 OR Karnofsky 60-100%
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3;
  * Platelet count >= 100,000/mm3;
  * White Blood Count (WBC) >= 3,000/mm3
* Hepatic:

  * aspartate aminotransferase-alanine aminotransferase (AST and ALT) =< 2.5 times upper limit of normal;
  * Bilirubin normal
* Renal:

  * Creatinine not elevated OR
  * Creatinine clearance >= 60 mL/min
* Cardiovascular:

  * No symptomatic congestive heart failure;
  * No unstable angina pectoris;
  * No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to decitabine
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior cytotoxic chemotherapy for thyroid cancer
* At least 6 months since prior external beam radiotherapy administered for locoregional disease in the thyroid bed or to the cervical or upper mediastinal lymph node regions (no more than 6,000 cGy)
* More than 6 months since other prior radiotherapy and recovered
* More than 6 months since prior therapeutic 131I > 10 mCi
* More than 18 months since prior cumulative 131I activity of at least 500 mCi
* More than 12 months since prior amiodarone (Unless 24-hour urinary iodine excretion is =< 500 mcg)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* More than 6 months since prior intrathecal iodinated contrast (Unless 24-hour urinary iodine excretion is =< 500 mcg)
* More than 3 months since prior IV or oral iodinated contrast for radiographic studies (Unless 24-hour urinary iodine excretion is =< 500 mcg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sherman, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Colorado at Denver, Aurora, Colorado
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consented at the University of Texas (UT) MD Anderson Cancer Center between 8/20/2004 and 4/28/2008. The trial was closed to new patient entry on 8/15/2008.
Groups:
- Treatment: Decitabine intravenous (IV) over 1 hour on days 1-5 and 8-12 of weeks 1 and 2 (course 1). Week 3, Iodine I 131 (131I) scanning using thyrotropin alfa injections. Participants whose scan do not demonstrate iodine uptake continue suppressive thyroid hormone therapy but no further study therapy; these participants who do show uptake undergo thyroid hormone withdrawal on weeks 4-8 and second course of decitabine (as in course 1) on weeks 7 and 8, with 131I therapy on week 9.
  Decitabine: Starting dose 6 mg/m^2 intravenously over 1 hour every day for 5 successive days for 2 weeks (10 doses), with possible second course.
  Iodine I 131: Undergo thyrotropin-alfa stimulated radioactive iodine scan
  Recombinant thyrotropin alfa: Undergo thyrotropin-alfa stimulated radioactive iodine scan
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of therapy.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Restoration of Radioiodine Uptake in Metastatic Lesions as Demonstrated by Diagnostic Whole-body Scanning After Decitabine Administration
Description: Number of participants with restoration of radioiodine responsiveness as determined by visible uptake on radioiodine scan in radiographically detectable metastatic foci of papillary or follicular thyroid carcinoma. Response to Decitabine defined as demonstration of radioiodine uptake determined by centralized blinded review of diagnostic scan. All who demonstrated radioiodine uptake in metastatic foci following decitabine therapy would then undergo thyroid hormone withdrawal and a second course of decitabine in preparation for therapeutic administration of radioiodine.
  Diagnostic radioiodine scans following decitabine therapy (week 3) with a radioiodine scan following thyrotropin alfa stimulation, 0.9 mg intramuscular (IM) injection 24 and 48 hours before administration of the 131I for imaging. Whole body scans (WBS) performed using a gamma camera.
Time Frame: Week 3 following 2 weeks of Decitabine therapy
Population: Per protocol, 1 participant interpreted by local treating investigator as responsive (increased radioiodine uptake on diagnostic scan after therapy), entered second decitabine treatment receiving radioiodine therapeutic dose. Subsequent central review of both scans for formal protocol response interpreted scans as negative for radioiodine uptake.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
participants | 0

2. Secondary Outcome: Frequency of Adverse Events According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Summary of Adverse Events (AEs) by Maximum Grade where Grade 1 AEs >20%, Grade 2 AEs >10%, all Grade 3, Grade 4 and Grade 5 reported.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants
  Grade 1, Nausea | 42
  Grade 1, Fatigue | 33
  Grade 1, Oral Mucositis | 25
  Grade 1, Pharyngolaryngeal pain | 25
  Grade 1, Decreased white blood cell | 25
  Grade 2, Fatigue | 25
  Grade 2, Decreased white blood cell | 25
  Grade 2, Neutrophil count decreased | 16
  Grade 2, Lymphocyte count decreased | 16
  Grade 3, Decreased white blood cell | 42
  Grade 3, Neutrophil count decreased | 25
  Grade 3, Febrile neutropenia | 8
  Grade 3, Infections | 8
  Grade 3, respiratory disorders | 8
  Grade 4, Decreased white blood cell | 58
  Grade 5 | 0

3. Secondary Outcome: Efficacy of Subsequent Radioiodine Therapy in Terms of CR/PR/SD of Any Radiographic Disease.
Description: Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 6 months
Population: No secondary endpoints were measured as no patient met the primary endpoint. These secondary endpoints would only have been assessed if a patient had met the primary endpoint, restoration of radioiodine uptake to justify radioiodine therapy.
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Fludeoxyglucose (FDG) Uptake Measured by Positron Emission Tomography in Metastatic Tumor Sites Before and After DNA-methyltransferase Inhibitor Therapy (Optional). No Secondary Endpoints Were Measured as no Patient Met the Primary Endpoint.
Time Frame: Baseline to 3 weeks
Population: as for outcome 3
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Efficacy of Subsequent Radioiodine Therapy in Terms of Complete Response (CR)/Partial Response (PR)/Stable Disease (SD) of Any Radiographic Disease
Description: as for outcome 3
Time Frame: 3 months
Population: as for outcome 3
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Efficacy of Subsequent Radioiodine Therapy in Terms of Change in Serum Thyroglobulin Level
Time Frame: 6 months
Population: as for outcome 3
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Efficacy of Subsequent Radioiodine Therapy in Terms of Change in Serum Thyroglobulin Level.These Secondary Endpoints Would Only Have Been Assessed if a Patient Had Met the Primary Endpoint, Restoration of Radioiodine Uptake to Justify Radioiodine Therapy.
Time Frame: 3 months
Population: as for outcome 3
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Routine clinical trial adverse event monitoring during study treatment for one month or up to six months total, depending on whether additional decitabine and radioactive iodine treatment received. Total study period 5/3/04 to 08/15/08.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Infection with Grade 3 or 4 neutrophils
White blood cell decreased (Blood and lymphatic system disorders) | 5 (5)
Neutrophil count decreased (Blood and lymphatic system disorders) | 9 (9)
Acute Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
Abdominal pain (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (General disorders) | 1 (1)
Chest wall pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (9)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Infections and infestations) | 3 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less